CLINICAL TRIAL: NCT04149743
Title: HEMOTAG® Assessment for Short-term Outcomes of Heart Failure [HATS-OFF]
Brief Title: HEMOTAG® Assessment for Short-term Outcomes of Heart Failure
Acronym: HATS-OFF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aventusoft, LLC. (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Cleveland Clinic Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 20192767/HT-17-VV-020; 1R44HL145941 (NIH)
Record Dates: First submitted 2019-10-29; First posted 2019-11-04 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure (HF)
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Randomized Standard of Care (No Intervention): Standard of Care
- Randomized Standard of Care with HEMOTAG (Active Comparator): Standard of Care with HEMOTAG
  Interventions: Diagnostic Test: Standard of Care with Hemotag

INTERVENTIONS:
Diagnostic Test: Standard of Care with Hemotag — Comparison of outcomes
  Other Names: Standard of Care
  Arms: Randomized Standard of Care with HEMOTAG

SUMMARY:
Evaluation of the HEMOTAG® system in a less controlled environment and concurrently develop the system for use by patients with heart failure.

DETAILED DESCRIPTION:
The overall objective of research is to test, adapt, refine and validate the HEMOTAG® system to be used outside the usual medical care environments to reduce hospital readmissions.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 22 years old.
* An index hospital admission for ADHF presenting with symptoms, clinical signs, and chest x-ray (CXR) findings of pulmonary congestion, receiving IV diuretics or vasoactive drugs and having a BNP > 350 or NT-pro BNP > 1800 pg/ml.
* Able to give informed consent.
* Participant's residence has adequate cellular data coverage.
* Participants with previous diagnosis of left ventricular ejection fraction (LVEF) <40% prior to the index hospitalization must have been treated for at least 90 days prior to enrollment with diuretics and beta-blocker (unless intolerant or contraindicated) and an ACE inhibitor or ARB or ARNi (unless intolerant or contraindicated).

Exclusion Criteria:

* Participants unable to provide informed, voluntary decision to participate in research study as determined by the investigator. (Exclude participants who necessitate the involvement of a legally authorized representative.)
* Terminal condition with life expectancy less than 6 months as determined by investigator.
* Participants with cardiac tamponade or constrictive pericarditis.
* Participants with left ventricular assistance device (LVAD device) or had a cardiac transplantation or listed for transplantation.
* Implantation of a CRT (cardiac resynchronization therapy) device during index hospitalization or intent to implant a CRT device.
* Presence of hemodynamically significant mitral and/or aortic valve disease, except mitral regurgitation secondary to left ventricular dilatation, as determined by investigator.
* Presence of hemodynamically significant obstructive lesions of left ventricular outflow tract, including aortic and sub-aortic stenosis, as determined by investigator.
* Severe primary pulmonary, renal or hepatic disease, as determined by investigator.
* Women of childbearing age (Age <50).
* History of pulmonary embolism of less than 3 months.
* Dialysis dependent or dialysis initiation expected within three months.
* Chronic home IV therapy or cardiac inotropes or diuretics.
* Physical deformity in the chest area or lesion that may prevent proper HEMOTAG application or adjustment.
* Illness/ Condition which may be aggravated or cause significant discomfort by the application of the HEMOTAG (skin issues, e.g. Intolerance to use of skin electrodes).
* Impaired cognitive ability or any other state that may prevent full compliance with the study protocol, according to investigator's assessment.
* Congenital heart malformations (Complex, or uncorrected congenital heart disease).
* Participant enrolled in another interventional study (observational or registries are not excluded).
* Participant HF is managed remotely with another monitoring device or program (for example: Pulmonary/ Lt Atrial pressure monitoring, lung fluid monitoring. BNP/pro-BNP or bioimpedance or ICD or biventricular pacemaker with impedance monitoring will be allowed unless it is part of another research protocol).
* Prisoners and wards of the state.
* Inability to provide informed consent (Must speak English or Spanish or Creole).

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The number of recurrent HF readmissions. [Monitoring period: 30 days] | 30 Days
  Determine if HEMOTAG can reduce the relative number of HF readmissions or ER visits versus standard of care. [Monitoring period: 30 days from time of participant's discharge from initial index hospitalization]

SECONDARY OUTCOMES:
Time from discharge until the first event of HF readmissions [Monitoring period: Event time assessed up to 3 months and 6 months from discharge. | 6 Months
  Time from discharge to the first event of HF readmissions or ER visits [Monitoring period:
  Event time assessed up to 3 months and 6 months from time of participant's discharge from initial study hospitalization.]
Number of total days lost to hospitalization due to HF events [Monitoring period: Expected average of 30 days, 3 months, 6 months] | 6 Months
  Total number of total days lost to hospitalization or ER visit due to HF events [Monitoring period: Expected average of 30 days, 3 months, 6 months from time of participant's discharge from index hospitalization.]
Time from discharge to all-cause mortality [Monitoring period: 30 days, 3 months,6 months] | 6 Months
  Time from discharge to all-cause mortality [Monitoring period: 30 days, 3 months,6 months from time of participant's discharge from initial study hospitalization.]
Skin irritation from HEMOTAG use [Time Frame: over the measurement period of 30 days] (Determine if subjects had skin irritation from use.) | 30 Days
  Incidence of skin irritation [Time Frame: over the measurement period of 30 days] (Determine if subjects had skin irritation from use of device.)

CONTACTS AND LOCATIONS:
Overall Officials: David Snipelisky, MD, Principal Investigator — Cleveland Clinic Florida
Locations (2):
- United States (2):
  - Cleveland Clinic Florida, Weston, Florida
  - Baylor Scott & White Research Institute, Temple, Texas

IPD SHARING:
Plan to Share IPD: No